CLINICAL TRIAL: NCT04928261
Title: A Single-arm, Multicentre, Pragmatic Trial Evaluating 6-months of HER2-targeted Therapy in Patients With HER2 Positive Early-stage Breast Cancer That Achieve a Pathological Complete Response to Neoadjuvant Systemic Therapy (REaCT-HER TIME)
Brief Title: Evaluating 6-months of HER2-targeted Therapy in Patients With HER2 Positive Early-stage Breast Cancer That Achieve a Pathological Complete Response to Neoadjuvant Systemic Therapy
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REaCT-HER TIME
Record Dates: First submitted 2021-05-04; First posted 2021-06-16 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: Cardiac toxicities; Her2 Positive; Pathological complete response
MeSH Terms: conditions — Breast Neoplasms; Cardiotoxicity | interventions — Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- De-escalated HER2 targeted treatment (Experimental): Patients with early-stage HER2-positive breast cancer who demonstrate a pathological complete response at time of surgery.
  Interventions: Drug: Trastuzumab

INTERVENTIONS:
Drug: Trastuzumab — Patients with early-stage HER2-positive breast cancer who demonstrate a pathological complete response at time of surgery will be treated with HER2 targeted therapy for a total of 9 treatments every 3 weeks (or its equivalent if given weekly) including the treatment received preoperatively.
  Other Names: Herceptin

SUMMARY:
The activity of trastuzumab in early-stage, HER2-positive breast cancer, has been demonstrated in many studies, with meta-analyses showing that in combination with a variety of chemotherapy backbones, trastuzumab reduces the risk of recurrence by nearly half, and death by a third. However, treatment with trastuzumab can result in cardiotoxicity, including heart failure, as well as the significant cost of treatment and the requirement for patients to attend the chemotherapy unit for treatment every 3 weeks for one year. Therefore there has been increasing interest in identifying which patients can safely have less treatment. The investigators therefore propose a real-world, single arm, multicentre trial evaluating 6 months of HER2 targeted therapy, for patients with early-stage, HER2 positive breast cancer, who achieve a pathological complete response (pCR) with upfront systemic chemotherapy and HER2 targeted therapy.

DETAILED DESCRIPTION:
The activity of trastuzumab in early-stage, HER2-positive breast cancer, has been demonstrated in many studies, with meta-analyses showing that in combination with a variety of chemotherapy backbones, trastuzumab reduces the risk of recurrence by nearly half, and death by a third. However, treatment with trastuzumab can result in cardiotoxicity, including heart failure, as well as the significant cost of treatment and the requirement for patients to attend the chemotherapy unit for treatment every 3 weeks for one year. Therefore there has been increasing interest in identifying which patients can safely have less treatment. The duration of adjuvant trastuzumab in early-stage breast cancer in the majority of studies was empirically set at 12 months, which became the de facto standard of care. Neoadjuvant treatment has become the new standard of care for patients with early-stage HER2-positive disease. While patients with residual disease benefit from further alternative treatment those with a pathological complete response (pCR) have an excellent outcome and are candidates for treatment de-escalation. The investigators therefore propose a real-world, single arm, multicentre trial evaluating 6 months of HER2 targeted therapy, for patients with early-stage, HER2 positive breast cancer, who achieve a pCR with upfront systemic chemotherapy and HER2 targeted therapy.

ELIGIBILITY:
Inclusion Criteria:

* Early-stage (I-III, i.e. non-metastatic) as per AJCC 8th edition, ER/PR positive or negative, HER2-positive as per 2018 American Society of Clinical Oncology/College of American Pathologists human epidermal growth factor receptor 2 (HER2) testing in breast cancer guidelines.
* Treated with neoadjuvant chemotherapy and HER2 targeted therapy preoperatively with a pathological complete response (pCR) defined as the absence of residual invasive cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy at surgery. Must have received less than 6 months of HER2 targeted therapy
* Able to provide verbal consent and complete questionnaires in English or French

Exclusion Criteria:

* Residual invasive disease following neoadjuvant therapy, or metastatic disease
* Contraindication to further HER2-targeted therapy following completion of neoadjuvant treatment
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the trial protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Multiple site activation | 1 year after first participant is accrued
  Evaluating the feasibility of multiple Canadian site activation within the first year of study accrual. Achieved by the activation of at least 4 Canadian sites within 1 year of the first patient being accrued into the study.
Medical oncologist active participation | Through to end of accrual - average 2 years
  Evaluating the number of medical oncologists at each study site who actively participate in the trial. Active participation includes approaching eligible patients for the study, as well as following up with the patients who are taking part in the study.
Enrolment of at least 50 participants across all sites within 9 months of the fourth site accruing its first participant | 9 months after fourth site accrues first participant
  Enrolment of at least 50 participants across all sites within 9 months of the fourth site accruing its first participant.

SECONDARY OUTCOMES:
Cardiac events | 3 years after study enrolment
  Cardiac events defined as death from a cardiac or heart failure of New York Heart Association (NYHA) class III or IV, or with a decrease in the left ventricular ejection fraction of at least 10 percentage points from baseline to a value of less than 50%. Cardiac monitoring will be assessed as per physician standards
Rate of HER2-positive treatment discontinuation | 6 months after study enrolment
  De-escalated HER2-positive treatment discontinuation and the reasons why treatment was discontinued
Health-related quality of life | Baseline, 3, 6, 12 and 36 months after study enrolment
  Health-related quality of life measure using the EuroQol-5 Dimension-5 Level (EQ-5D-5L) questionnaire.
Incremental cost-effectiveness ratios | 3 years from study enrolment
  The difference in cost between 6 months of HER2-positive therapy versus the standard 12 months of HER2-positive therapy.
Disease free survival | 3 years from study enrolment
  Disease Free Survival (DFS), defined as the percentage of people in the trial who are alive and disease-free (no local invasive breast cancer recurrence, new local invasive breast cancer) at 3 years
Overall survival | 3 years from study enrolment
  Overall Survival (OS), defined as the number of people alive, with or without signs of cancer at 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Sharon McGee, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital Cancer Centre, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Bradbury M, Savard MF, Vandermeer L, Clemons L, Pond G, Hilton J, Clemons M, McGee S. Shorter Durations of Anti-HER2 Therapy for Patients with Early-Stage, HER2-Positive Breast Cancer: The Physician Perspective. Curr Oncol. 2023 Dec 14;30(12):10477-10487. doi: 10.3390/curroncol30120763. PMID 38132397
- See also: The Rethinking Clinical Trials (REaCT) website — https://react.ohri.ca/